CLINICAL TRIAL: NCT03002441
Title: Same-day Cervical Preparation With Dilapan-S™ Plus Buccal Misoprostol Compared to Overnight Dilapan-S™ Before Dilation and Evacuation at 16 to 20 Weeks' Gestation: A Randomized Controlled Trial
Brief Title: Same-day Cervical Preparation Before Dilation and Evacuation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Planned Parenthood of Greater New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Same Day CPrep
Record Dates: First submitted 2016-12-06; First posted 2016-12-23 (Estimated); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Cervical Dilation Prior to Dilation and Evacuation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Same-day Dilators (Active Comparator): Participants will have Dilapan-S cervical dilators placed 4-6 hours prior to D&E and will receive 400 mcg buccal misoprostol pills 3 hours prior to D&E.
  Interventions: Device: Same-Day Dilapan-S
- Overnight dilators (Active Comparator): Participants will have Dilapan-S cervical dilators placed the day prior to their D&E procedure and will receive buccal placebo pills (vitamin B12) 3 hours prior to D&E.
  Interventions: Device: Overnight Dilapan-S

INTERVENTIONS:
Device: Same-Day Dilapan-S — Dilapan-S cervical dilators placed the same day as the D&E procedure
  Arms: Same-day Dilators
Device: Overnight Dilapan-S — Dilapan-S cervical dilators placed the day prior to D&E procedure
  Arms: Overnight dilators

SUMMARY:
The purpose of this randomized trial is to compare same-day cervical preparation using Dilapan-S™ plus buccal misoprostol to overnight cervical preparation using Dilapan-S™ before D&E at 16.0 to 20.0 weeks.

Primary objective: To compare D&E operative time. We hypothesize that same-day Dilapan-S™ plus buccal misoprostol is non-inferior to overnight Dilapan-S™ with respect to operative time.

Secondary objectives: To compare treatment groups for the following: Pre-operative cervical dilation; need for mechanical dilation and ease of dilation if required; ability to complete D&E without further cervical preparation; ease of D&E; complications; pain; side effects; patient and provider satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Seeking pregnancy termination from 16 0/7 to 19 6/7 weeks of gestation on the day of enrollment.
* Eligible for pregnancy termination at PPNYC
* Able to give informed consent
* English speaking

Exclusion Criteria:

* Active bleeding or hemodynamically unstable at enrollment
* Signs of chorioamnionitis or clinical infection at enrollment
* Signs of spontaneous labor or cervical insufficiency at enrollment
* Spontaneous intrauterine fetal demise
* Allergy to Dilapan-S™ or misoprostol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Operative time | From initiation of D&E procedure to completion of D&E procedure, Study Day 2

CONTACTS AND LOCATIONS:
Overall Officials: Ila Dayananda, Principal Investigator — Planned Parenthood of Greater New York
Locations (1):
- Planned Parenthood of Greater New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim CS, Dragoman M, Porsch L, Markowitz J, Lunde B, Stoffels G, Dayananda I. Same-Day Compared With Overnight Cervical Preparation Before Dilation and Evacuation Between 16 and 19 6/7 Weeks of Gestation: A Randomized Controlled Trial. Obstet Gynecol. 2022 Jun 1;139(6):1141-1144. doi: 10.1097/AOG.0000000000004790. Epub 2022 May 2. PMID 35675611